CLINICAL TRIAL: NCT07039149
Title: Dual Antiplatelet Agents Therapy in the Emergency Department for Acute Coronary Syndrome (The DATES Study).
Brief Title: Pretreatment of Acute Coronary Syndrome With Dual Antiplatelet Agents
Acronym: DATES
Status: Recruiting | Type: Observational
Sponsor: Jordan Collaborating Cardiology Group (Other)
Responsible Party: Principal Investigator, Ayman J Hammoudeh, MD, FACC, Director, Department of Clinical Research; Director, Department of Internal Medicine, Jordan Collaborating Cardiology Group
Other Study IDs: DATES.2.25/irbIH1725
Record Dates: First submitted 2025-06-18; First posted 2025-06-26 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Major Bleeding; Major Adverse Cardiovascular and Cerebrovascular Events (MACCE)
Keywords: Dual antiplatelet therapy; Pretreatment with DAPT; Acute coronary syndrome
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult patients admitted for acute coronary syndrome via the ED: Patients with ACS presenting to the ED with a planned coronary angiography for possible coronary revascularization who get aspirin in the ED will be evaluated for bleeding and major cardiovascular events when they receive a second antiplatelet agent in the ED compared with in the cath lab.

SUMMARY:
This is a chart review of data on use of antiplatelet (AP) medications for acute coronary syndrome in the ER. Guidelines recommend giving aspirin in the ER and a second AP agent in the cath lab. What is the outcome when the 2 agents are given n the ER?

DETAILED DESCRIPTION:
Dual antiplatelet therapy (DAPT) is a standard treatment in ST-elevation myocardial infarction (STEMI) and non-ST-segment-elevation acute coronary syndrome (NSTEACS) . However, the timing of initiation of DAPT in the Emergency Department (ED) has been defined by recent western guidelines (i.e., aspirin in the ER and and a second AP agent when the coronary anatomy has been denied in the cath lab. This strategy aims at decreasing the incidence of bleeding events. However, patients with ACS in the Middle East are younger than those in the West and have lower bleeding risk. The purpose of this study is to evaluate the incidence of major bleeding in patients who received DAPT in the ED according to the discretion of the treating physician.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Presenting with acute coronary syndrome (ST segment elevation myocardial infarction, non ST segment elevation myocardial infarction, and unstable angina).
* Antiplatelet medication (s) prescribed during index admission to hospital.
* Willingness of the patient to be called for follow up up to 1 year after index hospitalization.

Exclusion Criteria:

* Non cardiac chest pain.
* No administration of antiplatelet agents during hospitalization.
* Refusal of contact for follow up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will enroll adult patients, men and women, who present to the emergency department (ED) with acute coronary syndrome (ST segment elevation myocardial infarction, non ST segment elevation myocardial infarction, and unstable angina) and who are prescribed aspirin in the ED and a second oral antiplatelet medication either in the ED (not according to recent guidelines) or upon identification of the coronary anatomy in the cath lab (based on recent guidelines). Incidence of bleeding and other cardiovascular events in these patients based in timing of administering the antiplatelet therapy.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Major bleeding event | From enrollment to the end of the study at 1 year.
  Major bleeding event is defined as any of the following: 1. bleeding causing hemodynamic compromise, 2. bleeding necessitating blood transfusion, or 3. bleeding in a closed space (intracerebral intraspinal and intraocular).

SECONDARY OUTCOMES:
Major adverse cardiovascular and cerebral events | from enrollment to 1 year
  Occurrence of any of the followings: 1. Cardiovascular death (death due to documented cardiovascular event: fatal myocardial infarction, or fatal stroke), 2. Non fatal myocardial infarction (two of three criteria: ischemic chest pain, electrocardiographic changes [ST segment deviation and T wave inversion] and elevated cardiac enzymes), 2. Definite stent thrombosis (demonstrating a thrombus in the stent on coronary angiography), 3. Non fatal stroke (new neurological deficit compatible with cerebral ischemia, brain imaging by computed tomography or magnetic resonance showing typical stroke, ischemic or hemorrhagic), 4. Coronary revascularization by percutaneous intervention or coronary bypass surgery.

CONTACTS AND LOCATIONS:
Locations (2):
- Jordan (2):
  - Jordan University Hospital, Amman
  - Istishari Hospital, Amman

IPD SHARING:
Plan to Share IPD: Undecided